CLINICAL TRIAL: NCT01385657
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential Ascending, Repeated-Dose Study of the Safety, Tolerability, and Pharmacokinetics of Subcutaneous REGN668 in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Safety and Tolerability of Dupilumab in Participants With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-AD-1026
Record Dates: First submitted 2011-06-09; First posted 2011-06-30 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Experimental): Placebo (for Dupilumab) as a single subcutaneous (SC) injection on Day 1, 8, 15, and 22
  Interventions: Drug: Placebo; Other: Background treatment
- Dupilumab 150 mg (Experimental): Dupilumab 150 mg as a single SC injection on Day 1, 8, 15, and 22
  Interventions: Drug: Dupilumab; Other: Background treatment
- Dupilumab 300 mg (Experimental): Dupilumab 300 mg as a single SC injection on Day 1, 8, 15, and 22
  Interventions: Drug: Dupilumab; Other: Background treatment

INTERVENTIONS:
Drug: Placebo — A total of 4 doses were administered.
  Arms: Placebo
Drug: Dupilumab — A total of 4 doses were administered.
  Other Names: REGN668; SAR231893; Dupixent
  Arms: Dupilumab 150 mg; Dupilumab 300 mg
Other: Background treatment — Participants were required to apply stable doses of an additive-free, basic bland emollient on the affected areas of the skin twice daily throughout the study.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of repeated subcutaneous (SC) doses of Dupilumab in participants with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years or older;
2. Chronic AD diagnosed by the Eichenfield revised criteria of Hannifin and Rajka that had been present for at least 3 years before the screening visit;
3. Eczema Area and Severity Index (EASI) score ≥ 12 at the screening and baseline visits;
4. Investigator's Global Assessment (IGA) score ≥ 3 at the screening and baseline visits;
5. ≥ 10% body surface area (BSA) of AD involvement at the screening and baseline visits;
6. History of inadequate response to a stable (≥ 1 month) regimen of topical corticosteroids or calcineurin inhibitors as treatment for AD within 3 months before the screening visit.

Exclusion Criteria:

1. Positive Hepatitis B surface antigen, and/or positive Hepatitis C antibody at the screening visit;
2. Treatment with an investigational drug within 8 weeks or within 5 half-lives, if known, whichever is longer, before the baseline visit;
3. Treatment with leukotriene inhibitors within 4 weeks before the baseline visit;
4. Treatment with systemic corticosteroids within 4 weeks before the baseline visit;
5. Treatment with topical corticosteroids, tacrolimus, and/or pimecrolimus within 1 week before the baseline visit;
6. Systemic treatment for AD with an immunosuppressive/immunomodulating substance within 4 weeks before the baseline visit;
7. Chronic or acute infection requiring treatment with oral or IV antibiotics, antivirals, or antifungals within 4 weeks before the screening visit or superficial skin infections within 1 week before the screening visit;
8. Known history of human immunodeficiency virus (HIV) infection;
9. History of clinical parasite infection, other than treated trichomoniasis;
10. History of malignancy within 5 years before the baseline visit, with the following exceptions: participants with a history of completely treated carcinoma in-situ of cervix, and non-metastatic squamous or basal cell carcinoma of the skin were allowed;
11. Any medical or psychiatric condition which, in the opinion of the investigator or the sponsor's medical monitor, would place the participant at risk, interfere with participation in the study, or interfere with the interpretation of study results;
12. Pregnant or breast-feeding women;
13. Unwilling to use adequate birth control, if of reproductive potential and sexually active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-07-31 (Actual); Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) | Baseline up to end of study (up to Day 85)
  An adverse event (AE) was defined as any untoward medical occurrence in a participant who received investigational medicinal product (IMP) without regard to possibility of causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a study drug, whether or not considered related to the study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was considered as medically important event. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to the end of study visit [Day 85]). Any TEAE included participants with both serious and non-serious AEs.

SECONDARY OUTCOMES:
Pharmacokinetics of Dupilumab: Peak Plasma Concentration (Cmax) | Day 22 (pre-dose), 25, 29, 36, 43, 50, 57, 64, 71 and Day 85
  Maximum Plasma Concentration of functional Dupilumab observed following the fourth (last) dose.
Pharmacokinetics of Dupilumab: Last Positive (Quantifiable) Concentration (Clast) | Day 22 (pre-dose), 25, 29, 36, 43, 50, 57, 64, 71 and Day 85
  Last Positive (Quantifiable) Concentration of Dupilumab.
Pharmacokinetics of Dupilumab: Time of the Last Positive (Quantifiable) Concentration (Tlast) | Day 22 (pre-dose), 25, 29, 36, 43, 50, 57, 64, 71 and Day 85
  Mean time of last measurable concentration of Dupilumab in actual days.

OTHER OUTCOMES:
Percentage of Participants with Investigator's Global Assessment (IGA) Score of "0" or "1" at Day 29/ Week 4 (End of Treatment Period) | At Day 29/ Week 4
  IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score of "0" or "1" at Week 4 are reported.
Percent Change From Baseline in Body Surface Area (BSA) Affected by Atopic Dermatitis to Week 4 | Baseline to Day 29/ Week 4
  BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score to Week 4 | Baseline to Day 29/ Week 4
  The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score at Week 4 | Baseline to Day 29/ Week 4
  SCORAD was a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Percent Change From Baseline in 5-D Pruritus Scale to Week 4 | Baseline to Day 29/ Week 4
  The 5-D Pruritus was a 5-question tool used in clinical trials to assess 5 dimensions of background itch: degree, duration, direction, disability, and distribution. Each question corresponded to 1 of the 5 dimensions of itch. Participants rated their symptoms over the preceding 2-week period on a scale of 1 (least affected) to 5 (most affected). Total score ranges from 1 (least affected) to 25 (most affected).
Change From Baseline in Average Weekly Pruritus Numerical Rating Scale (NRS) Score to Week 4 | Baseline to Day 29/ Week 4
  Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (12):
- Australia (4):
  - Kogarah, New South Wales
  - Woolloongabba, Queensland
  - Carlton, Victoria
  - Nedlands, Western Australia
- Germany (5):
  - Hanover, Lower Saxony
  - Bonn, North Rhine-Westphalia
  - Berlin
  - Gera
  - Münster
- New Zealand (3):
  - Sydenham, Christchurch
  - Caversham, Dunedin
  - Auckland

REFERENCES:
- [Result] Hamilton JD, Suarez-Farinas M, Dhingra N, Cardinale I, Li X, Kostic A, Ming JE, Radin AR, Krueger JG, Graham N, Yancopoulos GD, Pirozzi G, Guttman-Yassky E. Dupilumab improves the molecular signature in skin of patients with moderate-to-severe atopic dermatitis. J Allergy Clin Immunol. 2014 Dec;134(6):1293-1300. doi: 10.1016/j.jaci.2014.10.013. PMID 25482871
- [Result] Beck LA, Thaci D, Hamilton JD, Graham NM, Bieber T, Rocklin R, Ming JE, Ren H, Kao R, Simpson E, Ardeleanu M, Weinstein SP, Pirozzi G, Guttman-Yassky E, Suarez-Farinas M, Hager MD, Stahl N, Yancopoulos GD, Radin AR. Dupilumab treatment in adults with moderate-to-severe atopic dermatitis. N Engl J Med. 2014 Jul 10;371(2):130-9. doi: 10.1056/NEJMoa1314768. PMID 25006719